CLINICAL TRIAL: NCT06415201
Title: Scenario-based Clinical Interview Data Construction and User Experience Evaluation
Brief Title: Interactive AI-based Mental Health Service for the Patients With Cancer
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Dongguk University Medical Center (Unknown); Eulji University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HI23C0315
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-10

CONDITIONS: Cancer
Keywords: mental health; distress; interactive artificial intelligence; virtual human
MeSH Terms: conditions — Neoplasms; Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Survey of unmet medical needs: 20 people
- User experience evaluation: 40 people
  Interventions: Other: Interactive Artificial Intelligence
- Clinical interview data collection: 200 people

INTERVENTIONS:
Other: Interactive Artificial Intelligence — scenario based AI to assess, classify, explain and conduct supportive interviews
  Groups: User experience evaluation

SUMMARY:
The aims of this study are developments of mental health care services for cancer patients based on interactive artificial intelligence. To do these things, survey of unmet medical needs and data collection of clinical interviews will be done, and newly developed assessment and intervention scenarios will be simulated to cancer patients group.

DETAILED DESCRIPTION:
A total of 20 people will be recruited from 3 institutions to investigate unmet medical needs. Based on the needs, we will develop scenarios to assess, classify, explain and conduct supportive interviews. We plan to develop a stress self-management scenario that helps manage lifestyle habits and provides meditation-based cognitive therapy. For moderate to severe distress, we plan to develop scenarios to link medical care and manage suicide risk. We plan to conduct interviews with a total of 300 people to collect clinical interview data for scenario development.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with malignant tumor and undergoing treatment, or patients undergoing follow-up after completing curative treatment

Exclusion Criteria:

* Patients unable to consent to research or be interviewed due to cognitive decline

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients without severe cognitive decline
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Distress | baseline
  Distress Thermometer
Quality of life measurement | baseline
  The world health organization quality of life (WHOQOL)
Stress | baseline
  Perceived Stress Scale (PSS-10)
Self-esteem | baseline
  Korean version of Rosenberg Self-Esteem Scale (K-RES)
Acceptance of Disability | baseline
  Acceptance of Disability Scale
Pain measurement | baseline
  PBPI (Pain belief & Perception inventory)
Insomnia | baseline
  ISI (Insomnia Severity Index)
Quality of sleep | baseline
  PSQI (Pittsburgh Sleep Quality Index)
Fatigue | baseline
  Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue)
Anxiety & Depression | baseline
  HADS (Hospital anxiety and depression scale)
Fear of Disease Progression | baseline
  FOP-SF (Fear of Disease Progression Short Form)
Social Support | baseline
  MOS Social support Survey

CONTACTS AND LOCATIONS:
Overall Officials: Bong-jin Hahm, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea